CLINICAL TRIAL: NCT05419024
Title: Imaging and Biopsy of People With HIV-1 Undergoing Analytic Treatment Interruption
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 10000277; 000277-C
Record Dates: First submitted 2022-06-11; First posted 2022-06-15 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-08-13

CONDITIONS: HIV
Keywords: Human Immunodeficiency Virus; Antiretroviral Therapy; FDG-PET; Reservoir
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATI (Experimental): Participants randomized to ATI will halt their ART medications starting 2 weeks (more or less 3 days) after the first imaging visit. This plan will be discussed with participants during the baseline visit. Patients will be contacted 1-3 days prior to ATI initiation. ATI may be delayed or cancelled if there are new safety concerns. HIV plasma viral levels and CD4 counts will be monitored every week during the ATI phase. If a participant meets any of the ART restart criteria during the ATI phase, then they will discontinue ATI and restart ART. Participants who do not meet restart criteria will remain off ART and continue to be monitored weekly until they have been on ATI for 90 days, and then will restart ART.
  Interventions: Other: Acute Treatment Interruption
- Continue ART (No Intervention): Participants will continue on their pre-study ART throughout the trial.

INTERVENTIONS:
Other: Acute Treatment Interruption — Participants randomized to ATI will halt their ART medications starting 2 weeks (more or less 3 days) after the first imaging visit. This plan will be discussed with participants during the baseline visit. Patients will be contacted 1-3 days prior to ATI initiation. ATI may be delayed or cancelled if there are new safety concerns. HIV plasma viral levels and CD4 counts will be monitored every week during the ATI phase. If a participant meets any of the ART restart criteria during the ATI phase, then they will discontinue ATI and restart ART. Participants who do not meet restart criteria will remain off ART and continue to be monitored weekly until they have been on ATI for 90 days, and then will restart ART.
  Arms: ATI

SUMMARY:
Background:

Human immunodeficiency virus (HIV) infects CD4 T cells. There is no cure for HIV. People with HIV need to take daily medications called antiretroviral therapy (ART) to control their infection. ART stops HIV from infecting cells, but HIV does not go away. Some infected cells remain. If ART is stopped, then HIV levels will rise and infect more cells.

Objective:

To compare changes in the amount of virus in blood and lymph nodes after a short treatment interruption.

Eligibility:

Adults aged 18 years or older who are undergoing ART for HIV infection.

Design:

Participants will be screened with a physical exam, including blood tests. They will be assigned to 1 of 2 groups:

One group will stay on ART. They will have 2 study visits: the first 45 days after screening, and the second 12 to 16 weeks later. They will have a PET/CT scan at each visit. A substance called a tracer will be injected into their arm. They will lie still on a table that moves through a doughnut-shaped machine. This process takes up to 2 hours.

The other group will stop ART for no more than 90 days. This group will have 3 PET/CT scans over 8 months. Once they stop ART, they will visit the clinic weekly for blood tests. After restarting ART, they will continue to visit the clinic weekly until their HIV level is safe.

All participants will have small samples of tissue taken from lymph nodes. They may also opt to provide semen samples or vaginal fluid. They may have samples taken of bone marrow or the fluid inside their spinal column.

DETAILED DESCRIPTION:
Study Description:

HIV persistence during antiretroviral therapy (ART) is the principal obstacle preventing cure, and new studies are essential to understand mechanisms and sources of persistence. Analytic treatment interruption (ATI) studies provide opportunities for detailed evaluation of mechanisms underlying HIV persistence and viral rebound, and can be especially useful in characterizing early events in HIV reactivation. Early viral dynamics of rebound have not been extensively characterized however, in part because commercial assays for HIV viremia are relatively insensitive for changes in low levels of HIV RNA. Assays with single copy sensitivity, such as the HIV Molecular Monitoring Core gag (HMMC gag) assay are > 100-fold more sensitive than commercial assays, thus increasing sensitivity for detecting change in HIV RNA levels in plasma. HMMC gag is also useful in quantifying HIV in cellular sites of persistence such as lymphoid tissues during early rebound. The use of more sensitive assays will permit characterization of events in early rebound. Studies of early rebound will facilitate investigation of immune and other correlates of rebound viremia. One potential correlate of rebound is increased metabolic activity resulting from increases in HIV production, or changes in the inflammatory milieu or both. Metabolic activity can be detected by 18fluorodeoxyglucose (FDG) positron emission tomography (PET). Investigating the dynamics of HIV rebound, inflammation, and metabolic activation will shed new light on mechanisms of persistence and rebound. We hypothesize that within 10 days of ATI, viral nucleic acid levels will increase in blood or lymphoid tissue. To investigate this hypothesis, we will perform a detailed study of HIV dynamics and metabolic imaging during ATI. Participants undergoing long term ART will undergo FDG PET imaging to identify areas of high and low metabolic uptake in lymphoid tissue after being randomized 1:1 to either continue ART or to ATI. Tissue samples will be collected by biopsy from areas of high and low FDG uptake. In participants randomized to ATI, blood collection, FDGPET and lymph node biopsy will be repeated 10 days after discontinuing ART. ATI will be continued until specific ART restart criteria are achieved, or a maximum of 90 days of ATI, and specimen collection will take place after viral suppression is re-achieved. Participants randomized to continue ART will have a second FDG-PET and specimen collection 12 to 16 weeks after the first collection. During the study, participants will undergo assessments of genetic characteristics of HIV populations (diversity, phylogenetics, and clonal structure) in plasma and lymphoid tissue. In addition to investigating HIV in plasma and lymphoid tissue, optional assessments of non-lymphoid anatomic compartments, including cerebrospinal fluid (CSF) obtained by lumbar puncture (LP), may be performed to evaluate characteristics of these anatomic compartments, which are known to be sources of HIV persistence.

Primary Objective:

Quantify the relative changes in blood HIV nucleic acids (RNA and DNA) and lymph node nucleic acids (RNA and DNA) from baseline to Day 10 (+/- 3 days) in the ATI vs no ATI arms.

Secondary Objectives:

1. Determine levels of 18F uptake in CT/PET imaging in individuals randomized to ATI vs no ATI
2. Characterize HIV populations (levels of HIV nucleic acids, genetic sequence of HIV genomes, integration sites of proviruses) in sampled tissues, peripheral blood mononuclear cells (PBMCs), and plasma prior to and following ATI, and after ART resumption.
3. Assess relationship between changes in 18F uptake and genetic characteristics (e.g., diversity, phylogenetics, and clonality) of HIV populations prior to, during, and after ATI.
4. Assess relationship between changes in soluble and cellular immune parameters and imaging findings during viral rebound.
5. Estimate replication competence of HIV variants from different anatomic compartments (sampled lymphoid tissues, PBMCs, plasma, semen, vaginal fluid, bone marrow and CSF).
6. Compare kinetics of viral rebound after ATI with changes in immune activation markers.

Tertiary/Exploratory Objectives:

1. Evaluate interaction of host characteristics, HIV population characteristics, and immune profiles.
2. Investigate HIV reactivation in other anatomic locations (CSF, semen, vaginal fluid, or bone marrow) in individuals who elect to undergo optional LP, semen or vaginal fluid collection, or bone marrow biopsy.
3. Evaluate the relationship between FDG-PET SUV and immunologic markers.
4. Investigate impact of ATI-associated changes in drug levels with changes in viral and immunologic characteristics.

Primary Endpoint:

Fold increase in HIV nucleic acids (RNA and DNA) in blood or lymphoid compartments from baseline to 10 day ATI vs baseline to no ATI

Secondary Endpoints:

1. Change in 18F uptake in individuals randomized to ATI vs no ATI.
2. Change in levels of HIV DNA, structure of HIV populations and integration site distribution to assess clonal distribution at different biopsy sites, semen, vaginal fluid, and PBMCs.
3. Correlation between regional and overall change in 18F with HIV DNA and RNA sequencing characteristics pre-ATI to post-ATI.
4. Cytokine and T-cell profiles during suppression and after ATI criteria for treatment resumption are met.
5. HIV RNA and DNA sequence analyses for genetic studies and potential for replication competence.
6. Correlation of HIV RNA levels and cytokine and T-cell profiles.

Tertiary/ExploratoryEndpoints:

1. Correlations between HIV population markers, lymphocyte phenotype parameters, and participant characteristics.
2. Comparative analysis of HIV DNA and RNA, levels of inflammatory markers, cytokine profiles, and antibody levels at different sites.
3. Correlation between regional and overall change in PET standardized uptake value (SUV) with changes in cytokine and T-cell profiles pre-ATI and post-ATI.
4. Correlations of viral population changes, HIV DNA levels, HIV RNA levels, and immune markers with drug levels.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants must meet all of the following criteria to be eligible for this study:

1. Aged >=18 years.
2. People with HIV-1 documented using US Food and Drug Administration-approved screening and confirmatory or supplemental assays in Centers for Disease Control and Prevention (CDC)-recommended testing strategies.
3. Established medical care outside NIH.
4. Able to provide informed consent.
5. Willing to allow samples to be stored for future research.
6. Willing to allow genetic testing.
7. Undergoing cART using recommended, alternative, or other regimens as defined by "Guidelines for the Use of Antiretroviral Agents in Adults and Adolescents with HIV."
8. Viral RNA <40 copies/mL plasma by conventional assay for at least 3 years (blips [transient increases within 6 weeks] of <200 copies/mL are allowable when succeeding viral levels return to <40 copies/mL on subsequent testing).
9. CD4 cell count >=350 cells/microliter.
10. Willing to interrupt ART for up to 90 days.
11. Willing to use a barrier method of contraception, such as condoms or dental dams, when engaging in sexual activity, or remain abstinent during ATI and after re-initiating ART until viral re-suppression is achieved, to prevent pregnancy and transmission of HIV.

EXCLUSION CRITERIA:

Participants who meet any of the following criteria will be excluded from this study:

1. Active intercurrent illness or infection, including fever >38 degrees Celsius.
2. Known history of initiating ART during the first year of infection with HIV. Participants will be considered to have initiated ART within 1 year of infection as defined by documented screening/confirmatory seroconversion (positive testing within one year of non-reactive HIV enzyme-linked immunosorbent assay).
3. Pregnant.
4. Breastfeeding.
5. Currently undergoing therapy with drugs that, in the judgment of the investigators, may interfere with biodistribution of FDG, including prednisolone, valproate carbamazepine, phenytoin, phenobarbital, and catecholamines.
6. Undergoing ART that is incompatible with an ATI.
7. Has undergone PET/CT within the last 6 months.
8. History of poorly controlled diabetes that, in the judgement of the investigators, would prevent completion of PET/CT scan.
9. Vaccination within the previous 4 weeks.
10. History of ATI within the past 1 year.
11. Has comorbid illness for which, in the judgment of the investigators, an ATI will represent elevated risk.
12. Active opportunistic infection as defined by the Guidelines for the Prevention and Treatment of Opportunistic Infections in Adults and Adolescents with HIV.
13. Significant active substance abuse or psychiatric illness that may, in the judgment of the investigator, interfere with study visits or procedures.
14. Allergy to planned anesthetic agents that are expected to be used. For local anesthetics, this is lidocaine. For sedation, this is midazolam and fentanyl.
15. Currently undergoing chronic systemic steroid therapy (corticosteroid nasal spray or inhaler, topical steroid use, and hormone replacement are acceptable).
16. Contraindication to use of IV contrast.
17. History of developing keloids.
18. Renal impairment: HIV-related kidney disease or estimated glomerular filtration rate (eGFR) CKD-EPI equation <60 mL/min/1.73 m^2. For individuals undergoing therapy with cobicistat or integrase strand inhibitors, GFR may be estimated using cystatin C or creatinine.
19. Active or chronic hepatitis B virus infection, with detectable hepatitis B surface antigen, hepatitis B virus DNA, or both.
20. Active hepatitis C virus infection, with detectable virus RNA.
21. History of HIV-associated dementia or progressive multifocal leukoencephalopathy.
22. Documented ARV drug resistance that, in the judgment of the investigator, would pose a risk of virologic failure should additional mutations develop during the study.
23. History of cardiovascular event or at high risk of an event (e.g., atherosclerotic cardiovascular disease score >20%) by a currently accepted risk calculator such as the 2023 AHA Predicting Risk of Cardiovascular Disease Events (PREVENT) or the 2018 ASCVD Risk Estimator Plus.
24. History of AIDS-defining illness according to CDC criteria within the past 3 years.
25. Hepatic impairment: aminotransferase >2.5 x the upper limit of normal or documented history of cirrhosis.
26. Any condition that, in the judgment of the investigator, contraindicates participation in this study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Fold increase in HIV nucleic acids (RNA and DNA) in blood or lymphoid compartments from baseline to 10 day ATI vs baseline to no ATI. | Up to day 90
  Compare change in HIV DNA and RNA after 10 day ATI in peripheral circulation and lymphoid compartment.

SECONDARY OUTCOMES:
6. Correlation of HIV RNA levels and cytokine and T-cell profiles. | Up to Month 6
  Assess relationship between immune and inflammatory markers with viral load.
5. HIV RNA and DNA sequence analyses for genetic studies and potential for replication. | Up to Month 6
  Evaluate viral population characteristics including completeness of genome over the course of the study.
4. Cytokine and T-cell profiles during suppression and after ATI criteria for treatment resumption are met. | Up to Month 6
  Comparison of immune and inflammatory milieu at baseline and after re-suppression post ATI.
3. Correlation between regional and overall change in 18F uptake with HIV DNA and RNA sequencing characteristics pre-ATI to post ATI. | Up to Month 6
  Determine if the relationship between SUV and viral populations differs at baseline and follow up depending on ATI versus no ATI.
2. Change in levels of HIV DNA, structure of HIV populations, and integration site distribution to assess clonal distribution at different biopsy sites, semen, vaginal fluid, and PBMCs. And following ATI, and after ART resumption. | Up to Month 6
  Compare characteristics of viral populations in sampled anatomical sites between baseline and follow up.
1. Change in 18F uptake in individuals randomized to ATI vs no ATI. | Up to Month 6
  Difference in SUV between baseline and second PET scan.

CONTACTS AND LOCATIONS:
Overall Officials: Chuen-Yen C Lau, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
There are only a few patients are being studied in this protocol. Data sharing might make it easier to identify participants.

REFERENCES:
- [Background] Lau CY, Adan MA, Maldarelli F. Why the HIV Reservoir Never Runs Dry: Clonal Expansion and the Characteristics of HIV-Infected Cells Challenge Strategies to Cure and Control HIV Infection. Viruses. 2021 Dec 14;13(12):2512. doi: 10.3390/v13122512. PMID 34960781
- [Derived] Lau CY, Adan MA, Earhart J, Seamon C, Nguyen T, Savramis A, Adams L, Zipparo ME, Madeen E, Huik K, Grossman Z, Chimukangara B, Wulan WN, Millo C, Nath A, Smith BR, Ortega-Villa AM, Proschan M, Wood BJ, Hammoud DA, Maldarelli F. Imaging and biopsy of HIV-infected individuals undergoing analytic treatment interruption. Front Med (Lausanne). 2022 Aug 22;9:979756. doi: 10.3389/fmed.2022.979756. eCollection 2022. PMID 36072945
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000277-C.html